CLINICAL TRIAL: NCT01075555
Title: Randomized Phase III Trial Sorafenib-Pravastatin Versus Sorafenib Alone for the Palliative Treatment of Child-Pugh A Hepatocellular Carcinoma
Brief Title: Sorafenib Tosylate With or Without Pravastatin in Treating Patients With Liver Cancer and Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000666232; FFCD-PRODIGE-11; FFCD-0803; EUDRACT-2009-015785-64; EU-21005
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Pravastatin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sorafenib (Active Comparator): sorafenib
  Interventions: Drug: sorafenib tosylate
- sorafenib + pravastatine (Experimental): sorafenib + pravastatine
  Interventions: Drug: pravastatin sodium; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: pravastatin sodium
  Arms: sorafenib + pravastatine
Drug: sorafenib tosylate

SUMMARY:
RATIONALE: Sorafenib tosylate and pravastatin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib tosylate may also stop the growth of liver cancer by blocking blood flow to the tumor. It is not yet known whether sorafenib tosylate is more effective when given alone or together with pravastatin in treating patients with liver cancer and cirrhosis.

PURPOSE: This randomized phase III trial is studying sorafenib tosylate given together with pravastatin to see how well it works compared with giving sorafenib tosylate alone in treating patients with liver cancer and cirrhosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the effects of sorafenib tosylate and pravastatin versus sorafenib tosylate alone on overall survival of patients with hepatocellular carcinoma and Child-Pugh Class A cirrhosis.

Secondary

* To evaluate the effect of this regimen on progression-free survival, time to progression, time to treatment failure, and quality of life (QLQ-C30 and FACT hep) in these patients.
* To evaluate the benefit of on-site monitoring versus the centralized data management monitoring of these patients.
* To characterize polymorphisms to specify the haplotype diversity in these patients.
* To test both diagnostic and prognostic signatures by quantitative RT-PCR to determine if they can predict response to these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center, Cancer of the Liver Italian Program (CLIP) score (0 vs 1 vs 2-4), WHO performance status (0 vs 1 vs 2), portal vein thrombosis (presence vs absence), and extrahepatic metastases (presence vs absence). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral sorafenib tosylate twice daily on days 1-28 and oral pravastatin once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral sorafenib tosylate twice daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients complete quality-of-life questionnaires (QLQ-C30 and FACT) at baseline and then every 4 weeks during and after completion of study therapy.

Blood and tissue samples may be collected for laboratory analysis, including pharmacogenomic studies.

After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatocellular carcinoma (HCC), meeting 1 of the following criteria:

  * Histologically confirmed HCC
  * If histological proof can not be obtained (e.g., ascites, coagulation disorders), the diagnosis may be made in cases of cirrhosis according to the 2005 EASL/AASLD criteria by demonstration of a focal hepatic lesion > 10 mm, meeting 1 of the following criteria:

    * Hypervascular tumor < 2 cm by 2 dynamic-imaging techniques (e.g., spiral CT scan, MRI scan, or ultrasound with contrast medium)
    * Hypervascular tumor ≥ 2 cm by 1 dynamic-imaging technique (e.g., spiral CT scan, MRI scan, or ultrasound with contrast medium)
* No progressive disease following prior treatment
* Not eligible for curative treatment (i.e., transplantation, resection, or percutaneous destruction) or chemoembolization
* Cancer of the Liver Italian Program (CLIP) prognosis score 0 to 4
* Child-Pugh score A
* No extrahepatic disease threatening the short- or medium-term vital prognosis

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 12 weeks
* Transaminases ≤ 5 times upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No other cancerous pathology, except for carcinoma in situ of the cervix, superficial bladder tumors, treated basal cell carcinoma, or any other cancer treated curatively ≥ 3 years ago
* No cardiac insufficiency (NYHA class II or IV congestive heart failure), arterial hypertension, uncontrolled arrhythmia, or myocardial infarction within the past 6 months
* No digestive hemorrhage within the past month
* No major bleeding disorder

PRIOR CONCURRENT THERAPY:

* No prior or other concurrent statins
* No prior sorafenib tosylate

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2010-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2014

SECONDARY OUTCOMES:
Progression-free survival | 2014
Time to progression | 2014

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Jouve, Principal Investigator — Hopital Du Bocage; Jacques Denis, MD, Principal Investigator — Hopital Louise Michel
Locations (1):
- Hopital Du Bocage, Dijon, France

REFERENCES:
- [Background] Jouve JL, Lecomte T, Bouche O, Barbier E, Khemissa Akouz F, Riachi G, Nguyen Khac E, Ollivier-Hourmand I, Debette-Gratien M, Faroux R, Villing AL, Vergniol J, Ramee JF, Bronowicki JP, Seitz JF, Legoux JL, Denis J, Manfredi S, Phelip JM; PRODIGE-11 investigators/collaborators. Pravastatin combination with sorafenib does not improve survival in advanced hepatocellular carcinoma. J Hepatol. 2019 Sep;71(3):516-522. doi: 10.1016/j.jhep.2019.04.021. Epub 2019 May 22. PMID 31125576